CLINICAL TRIAL: NCT05280288
Title: Effect of the App Bone@BC Version 4.0 Under the Follow-up for Patients With Early Breast Cancer - a Non-inferiority 2-year Randomized Controlled Trial (The BELIEVE@BC -Better Life Even After Breast Cancer Study)
Brief Title: Effect of the App Bone@BC Version 4.0 Under the Follow-up for Patients With Early Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Peter Schwarz, professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BELIEVE@BC
Record Dates: First submitted 2022-01-18; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Early-stage Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group (Standard care) (No Intervention): No intervention. This arm will continue standard clinical practice consisting of clinical assessment regarding side effects and management under follow-up having usual care alone conducted by physicians and therefore not able to use the app Bone@BC in any versions (access denied).
- The intervention group (Experimental): Intervention: This arm will be assigned to the intervention which will be that the participants will be invited to become active users of the app Bone@BC version 4.0 combined with usual care alone.
  Interventions: Device: Bone@BC app

INTERVENTIONS:
Device: Bone@BC app — Participants in the intervention group will be asked to use the Bone@BC app daily it will take them 1-3 minutes to answer the daily questions in the app concerning symptoms and physical activity. They will have access to a Questionnaire Prompt List in the app Bone@BC.
  Arms: The intervention group

SUMMARY:
Background Worldwide, an increasing number of people are affected by cancer. Breast Cancer is one of the most common cancers worldwide. Patients with early non-metastatic breast cancer are a growing group of survivors. The reason for this is that there has been an opportunity for early diagnosis, as well as improved treatment options. Patients with early breast cancer often experience endocrine side-effects such as loss of bone, increased weight, high levels of adipokine, lipids resistance, and hypertension after chemotherapy and anti-estrogen treatment resulting in reduced Health-Related Quality of Life.

Aim The aim is to investigate whether a Bone@BC app version 4.0 compared to usual care alone improves self-efficacy and provides at least as good HRQoL.

Methods A Randomized Controlled Trial (RCT) to decide whether the use of ePROs combined with usual care alone during follow-up for postmenopausal patients with early non-metastatic breast cancer in aromatase inhibitors with endocrine side-effects can maintain Health-Related Quality of Life, improve patient empowerment and self-efficacy compared to usual care alone.

DETAILED DESCRIPTION:
Background Worldwide, an increasing number of people are affected by cancer. In 2018, 18.1 million people were diagnosed with new cancer with a mortality rate of 9.6 million (53%). Breast Cancer is one of the most common cancers worldwide and the most frequent cancer diagnosis in Danish women. On average 4,700 new cases are diagnosed in Denmark per year among a total population of 5.7 million citizens.

Women with early non-metastatic breast cancer often experience a treatment-related physical and psychological burden.

Empowering people with the confidence and information to look after themselves when they can and visit the General Practice when they need to, gives people greater control of their health and encourages healthy behaviors that help prevent ill health in the long term. In many cases, people can care for their minor illnesses, reducing the number of consultations and enabling healthcare professionals to focus on caring for higher-risk patients, such as those with co-morbidities, the very young and elderly, managing long-term conditions, and providing new services. Around one in five visits to the General Practice are made for social needs such as isolation, debt management, low mood, and anxiety. Patient-reported outcomes (PROs) have the potential to improve patient-clinician communication, symptom management, involvement, and quality of life. Electronic patient-reported outcomes (ePROs) can facilitate appropriate and continuous symptom monitoring reported by the patients. A systematic review from 2019 finds that mobile Health (mHealth) apps with interventions focusing on breast cancer survivorship showed a positive effect by promoting weight loss, improving the Health-Related Quality of Life, and decreasing stress but they find that future research is needed exploring the impact of mHealth apps on breast cancer survivors undergoing follow-up.

Aim The aim is to investigate whether a Bone@BC app version 4.0 compared to usual care alone improves self-efficacy and provides at least as good Health-Related Quality of Life.

Study design and methods A two-arm prospective randomized controlled trial. The study will be a one-site non-inferiority 2- year RCT study. A total of (n=120) participants will be randomized into the intervention group (IG) (n=60), these participants will be invited to become active users of the app Bone@BC version 4.0 combined with usual care alone. The control group (CG) (n=60), consists of participants following have usual care alone, and therefore not able to use the app Bone@BC in any versions (access denied).

Recruitment and procedures Following a consecutive sampling strategy, the participants (total (n=120), intervention group (IG) (n=60), control group (CG) (n=60) in the RCT study will be recruited from the Endocrinology Out-Clinic at Rigshospitalet, Denmark. Today the Endocrinology Out-Clinic at Rigshospitalet receives 4-8 referrals a week from the Department of Oncology at Rigshospitalet, Denmark ward to treatment for metabolic symptoms. The patients will be recruited by the principal investigator Trine Lund-Jacobsen (TLJ) or the endocrinology physicians. The identification of patients will be given to the principal investigator (TLJ) in case the patients are accepted to be contacted for further written and oral information about the project, letter for the subject's rights is handed out and then be provided for obtaining written consent from the patient. The first 120 women who give written consent to participate in 1-year interim analysis and then until total inclusion. The patients who regret or refuse to give consent to participate in the study will be registered and we will note the reason why the patients refuse or regret to participate in the study. After providing consent and reflection time, the participants will be randomized for even the control group (CG) or the intervention group (IG) by closed letters.

Analytic plan An interim analysis is performed after one year. Following correlations analysis will be performed: Total score self-efficacy (SES6G), total score patient empowerment (heiQ), total score depression and anxiety (HADS), total score physical activity (SGPALS), and HRQoL (EORTC QLQ-C30).

The primary outcome is HRQoL and differences in HRQoL between using an app Bone@BC and standard usual care alone will be evaluated by a multivariable linear regression model adjusting for age, baseline HRQoL, baseline HADS, and baseline self-efficacy. Correlation analysis will identify correlations between specific symptoms and HRQoL. Paired t-tests will be used to compare the means for the control group (CG) and the intervention group (IG) and p-values < 0.05 are considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Age 50-70 years
* Danish speaking
* Diagnosed with EBC, stage I-III
* Eligible to receive (neo-) adjuvant chemotherapy or adjuvant treatments
* Access to an E-mail address
* Access to smart mobile electronic devices connected to the internet
* Willingness to have the app installed on the smart mobile electronic devices
* Ability to work with the app

Exclusion Criteria:

* Prior malignancy
* Pre-existing type 2 diabetes or other metabolic diseases
* Withdrawn or not given a consent form

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Quality of life measured by the European Organization for Research and Treatment of Cancer Quality of Life | baseline (0 months), and every three weeks
  Health-related quality of life scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
  Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.

SECONDARY OUTCOMES:
Changes in symptoms of depression and anxiety measured by Hospital Anxiety and Depression Scale | baseline (0 months), 1 year, and 2 year
  The Hospital Anxiety and Depression scale is a 14-item scale with seven items each for anxiety and depression subscales. Scoring for each item ranges from zero to three. A subscale score >8 denotes anxiety or depression.
Changes in self-efficacy measured by Self-efficacy for managing chronic disease 6-item scale (SES6G) | baseline (0 months), and every six weeks
  The Self-efficacy for managing chronic disease 6 item scale is a 6 item scale. Scoring for each item ranges from zero to ten. A high scale score represents a high self-efficacy.
Changes in patient empowerment measured by The Health Education Impact Questionnaire. | baseline (0 months), 1 year, and 2 year
  The Health Education Impact Questionnaire i a 42 items questionnaire with a 4 point response scale (strongly disagree, disagree, agree and strongly agree). Higher values in the Health Education Impact Questionnaire scales indicate better status, except for Emotional distress, where higher values indicate higher distress.
Changes in physical activity measured by The Grimby Physical Activity Level Scale 4 item questionnaire. | baseline (0 months), and every three weeks
  The Grimby Physical Activity Level Scale 4 item questionnaire is a 4 items questionnaire with following response scale:
  I (Sedentary). Mainly sedentary or engaged in light physical activity less than 2 h per week (e.g., reading books, watching television, or going to the cinema).
  II (Light to moderate). Light-to-moderate physical activity 2-4 h per week (e.g., walking, cycling for pleasure, gardening, housework, light exercise).
  III (Regular moderate). Moderate physical activity more than 4 h per week, or more strenuous activities 2-4 h per week (e.g. brisk walking, fast bicycling, heavy gardening, or exercises that makes you short of breath).
  IV (Regular vigorous). More strenuous physical activities more than 4 h per week, or regular vigorous exercise (e.g. competitive sport) several times a week.
Changes in in app user measured by Open source web analytics application Matomo Analytics | 1 year and the 2 year
  In-app user analytics will be collected to track user behavior such as the number of app sessions measured by numbers, length of app sessions measured by time (hours and sec.), frequency of use measured in numbers, data app was first opened measured as the specific site, geographic place measured as country, how many pages measured as numbers, how long time on the pages measured as time (hours and sec.), bounce rate measured as numers, and returning for the first time measured as numbers.
Bone@BC app | From start of radomization until end of study 24 months
  Patient-reported outcome(s) from the app on the questions provided daily on Health-Related Quality of Life, late side-effects, symptoms and concerns perspectives, and level of Physical Activity in the app Bone@BC). The daily questions will be from the Eortc Library and will be analysed in percentages.

IPD SHARING:
Plan to Share IPD: No